CLINICAL TRIAL: NCT05422339
Title: Efficacy of Gamification in Enhancing User Engagement in Visual Mapping Assistive Technology
Brief Title: Efficacy of Gamification in Enhancing User Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MapHabit, Inc. (Industry)
Responsible Party: Principal Investigator, Stuart Zola, Chief Scientific Officer, MapHabit, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Gamification Study (NIH PH II)
Record Dates: First submitted 2022-06-07; First posted 2022-06-16 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease; Dementia; Gamification; Assistive Technology
Keywords: Alzheimer disease; Dementia; Caregiver burden; activities of daily living; Assistive technology
MeSH Terms: conditions — Alzheimer Disease; Dementia; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: The study will be a randomized controlled clinical trial, in which two conditions will be investigated: a control and experimental condition.
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistical analyses of all data will be carried out independently of investigators by a biostatistical resource department of an academic health center for validation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified Intervention (Experimental): This condition involved the implementation of an assistive technology software (the MapHabit system) with added gamification features into the daily care of the participants. The experimental condition received the version that incorporates gamified content and structure. Gamification involved receiving four new cognitive games each month. The cognitive games that were chosen for the current study followed game types observed to be prevalent in literature centered on serious games within dementia research. These games aim for cognitive stimulation in slowing down symptom acuity. Game design elements of positive reinforcement, problem-solving, progression, and visual cues were implemented into game content and software.
  Interventions: Device: The MapHabit system (MHS)
- Non-gamified Intervention (Active Comparator): This control condition acted as the active comparator to the experimental condition. The same assistive technology, the MapHabit system, will be given to a separate group of participants with mild to moderate stage of ADRD. The difference here will be that the software will be a version that does not include gamification features. The Control Group watched several 40 to 55-minute educational videos that were sent to the participants' devices each month. The content involved topics such as Happiness, Memory, Nutrition/Diet, and Mindfulness. The intent was to have the two groups engaged for about equal lengths of time in each of their respective interventions.
  Interventions: Device: The MapHabit system (MHS)

INTERVENTIONS:
Device: The MapHabit system (MHS) — The MapHabit System (MHS) is a commercially available visual mapping software application that utilize visual, audio, and text media to create step-by-step visual guides to assist individuals and their caregivers in structuring and accomplishing activities of daily living (ADLs). The goal of the application is to develop and facilitate habits and routines using structured visual and auditory stimuli that can be customized by the user and can include educational and lesson-based material in addition to ADLs. The application will be made available to families through compatible smartphones and tablets. Depending on the condition, participants will receive a specific version of the application. The experimental condition will receive the version that incorporates gamified content and structure.
  The MHS is a general wellness product and there is no regulatory oversight of the MapHabit System mapping functionality. This functionality is not a regulated medical device.

SUMMARY:
As part of Phase II of the NIH SBIR grant, the study will conduct a randomized controlled clinical trial in which the MapHabit system's gamification is investigated to determine whether the assistive technology facilitates user engagement and retention. Additionally, the study will examine if the gamified software improves the quality of life of persons with dementia and reduce the burden of the respective care partners. Participants will be individuals with Alzheimer's disease or related dementias in mild to moderate stage of cognitive impairment, accompanied by their respective primary care partner (i.e., primary familial caregiver). The study will be a randomized controlled clinical trial, in which two conditions will be investigated: 1) experimental condition in which MHS+Gamification is implemented into the daily care received by participants 2) control condition in which the MHS alone and separate engagement material is incorporated into the participant's daily care. Sample size goal will strive for a total of 40 individual-caregiver dyads, 20 in each condition. The study duration will be a 6-month intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individual diagnosed with Alzheimer's disease or other related dementia (ADRD) in their mild to moderate stage of impairment
* Participating caregiver of individual with dementia must be the primary caregiver
* Proficient in English

Exclusion Criteria:

* Individual not diagnosed with ADRD
* Participating caregiver of individual with dementia is NOT the primary caregiver
* Not proficient in English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Zola, Principal Investigator — MapHabit, Inc.
Locations (1):
- MapHabit, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to szola@maphabit.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Boatman F, Golden M, Jin J, Kim Y, Law S, Lu A, Merriam N, Zola S. Assistive technology: Visual mapping combined with mobile software can enhance quality of life and ability to carry out activities of daily living in individuals with impaired memory. Technol Health Care. 2020;28(2):121-128. doi: 10.3233/THC-191980. PMID 31796718
- [Background] Kelleher J, Zola S, Cui X, Chen S, Gerber C, Parker MW, Davis C, Law S, Golden M, Vaughan CP. Personalized Visual Mapping Assistive Technology to Improve Functional Ability in Persons With Dementia: Feasibility Cohort Study. JMIR Aging. 2021 Oct 19;4(4):e28165. doi: 10.2196/28165. PMID 34269690
- [Background] Parker MW, Davis C, White K, Johnson D, Golden M, Zola S. Reduced care burden and improved quality of life in African American family caregivers: Positive impact of personalized assistive technology. Technol Health Care. 2022;30(2):379-387. doi: 10.3233/THC-213049. PMID 34334439
- [Background] Montgomery B, Mammen C, Golden M. Using a Gamification Approach to Enhance Continued Use of Assistive Technology Intervention in Persons Living with Dementia. OBM Geriatrics 2025; 9(2): 311; doi:10.21926/obm.geriatr.2502311

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 participants were targeted in order to account for expected enrollment attrition. The 60 participant enrollment include only the persons living with dementia (PLWD). Each participant was accompanied by their primary caregiver in order to receive necessary assistance in fully engaging in the study. All enrollment numbers, data, and outcomes reflect the 60 PLWD only, and do not include their accompanied caregivers. The subjects were randomly assigned to one of two groups.
Groups:
- Gamified Intervention: Participants were persons with mild/moderate stage of ADRD. Each participant were enrolled with the presence of their primary care partner, who was required in the assistance of the engagement of the intervention and completion of assessments throughout the study. Only the participant's tracked and self-reported data contributed to data collection. Accompanying care partners needed to be in a direct care partner relationship with the participant, defined as a care partner who spends at least eight hours per week with the participant. This condition involved the implementation of an assistive technology software (the MapHabit system) with added gamification features into the daily care of the participants. The application was made available through tablets. The experimental condition received the version that incorporates gamified content and structure. Gamification involved receiving four new cognitive games each month. The cognitive games that were chosen for the current study followed game types observed to be prevalent in literature centered on serious games within dementia research. These games aim for cognitive stimulation in slowing down symptom acuity. Game design elements of positive reinforcement, problem-solving, progression, and visual cues were implemented into game content and software.
- Non-gamified Intervention: Each participant enrolled together with their primary care partner in the same fashion described in the Gamified Intervention arm. This control condition acted as the active comparator to the experimental condition. The same assistive technology, the MapHabit system, was given to individuals with mild to moderate ADRD and their caregivers. The difference here was that the software was a version that did not include gamification features. The Control Group watched several 40 to 55-minute educational videos that were sent to the participants' devices each month. The content involved topics such as Happiness, Memory, Nutrition/Diet, and Mindfulness. The intent was to have the two groups engaged for about equal lengths of time in each of their respective interventions.
Period: Overall Study
Arm/Group | Gamified Intervention | Non-gamified Intervention
Started | 30 | 30
Completed | 13 | 15
Not Completed | 17 | 15
Not completed — Withdrawal by Subject | 17 | 15

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected for caregivers of enrolled participants. As described in pre-assignment details in Result Participant Flow, the current study strictly enrolled persons living with dementia, while being accompanied by their primary caregiver for appropriate support in fully engaging in the study.
Groups:
- Gamified Intervention: Participants were persons with mild/moderate stage of Alzheimer's disease and related dementias (ADRD). Each participant was enrolled with the presence of their primary care partner, who was required for assistance in the engagement of the intervention and completion of assessments throughout the study. Only participants directly contributed to data collection. Accompanying care partners needed to be in a direct care partner relationship with the participant, defined as a care partner who spends at least eight hours per week with the participant. This condition involved the implementation of an assistive technology software (the MapHabit system) with added gamification features into the daily care of the participants. The experimental condition received the version that incorporates gamified content and structure. Gamification involved receiving four new cognitive games each month. The cognitive games that were chosen for the current study followed game types observed to be prevalent in literature centered on serious games within dementia research. These games aim for cognitive stimulation in slowing down symptom acuity. Game design elements of positive reinforcement, problem-solving, progression, and visual cues were implemented into game content and software.
- Non-gamified Intervention: Each participant enrolled together with their primary care partner in the same fashion described in Gamified Intervention. This control condition acted as the active comparator to the experimental condition. The same assistive technology, the MapHabit system, was given to individuals with mild to moderate ADRD and their caregivers. The difference here was that the software was a version that did not include gamification features. The Control Group watched several 40 to 55-minute educational videos that were sent to the participants' devices each month. The content involved topics such as Happiness, Memory, Nutrition/Diet, and Mindfulness. The intent was to have the two groups engaged for about equal lengths of time in each of their respective interventions.
- Total: Total of all reporting groups
Arm/Group | Gamified Intervention | Non-gamified Intervention | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Customized [Count of Participants; unit: Participants]
  Age (%): 31-40 years old | 0 | 1 | 1
  Age (%): 41-50 years old | 1 | 1 | 2
  Age (%): 51-60 years old | 2 | 1 | 3
  Age (%): 61-70 years old | 1 | 2 | 3
  Age (%): 71-80 years old | 5 | 4 | 9
  Age (%): 81-90 years old | 4 | 4 | 8
  Age (%): 91-100 years old | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in User Interaction and Engagement From Baseline to 6 Months
Description: Our internal analytics of the software can assess the user's interactions with the application by tracking user's map use count per month. By combining these data points, we can determine the average engagement for each participant and compare them between groups.
Time Frame: User engagement (i.e., map count) was collected daily for the total duration of 180 days/6 months of the subject's participation. Usage data was segmented and analyzed via monthly basis.
Measure: Median (Standard Deviation); unit: Uses per Month
Groups:
- Gamified Intervention: Participants were persons with mild/moderate stage of Alzheimer's disease and related dementias (ADRD). Each participant was enrolled with the presence of their primary care partner, who assisted in the engagement of the intervention and completion of assessments throughout the study. Only participants directly contributed to data collection. Accompanying care partners needed to be in a direct care partner relationship with the participant, defined as a care partner who spends at least eight hours per week with the participant. This condition involved the implementation of an assistive technology software (the MapHabit system) with added gamification features into the daily care of the participants. The experimental condition received the version that incorporates gamified content and structure. Gamification involved receiving four new cognitive games each month. The cognitive games that were chosen for the current study followed game types observed to be prevalent in literature centered on serious games within dementia research. These games aim for cognitive stimulation in slowing down symptom acuity. Game design elements of positive reinforcement, problem-solving, progression, and visual cues were implemented into game content and software.
Arm/Group | Gamified Intervention | Non-gamified Intervention
Number analyzed (Participants) | 13 | 15
Uses per Month
  Month 1 | 32 (29.9) | 60 (89.0)
  Month 2 | 7 (29.3) | 36 (79.2)
  Month 3 | 8 (21.3) | 2 (39.7)
  Month 4 | 5 (13.2) | 4 (45.8)
  Month 5 | 4 (9.0) | 3 (38.7)
  Month 6 | 0 (16.0) | 4 (25.4)

2. Primary Outcome: Quality of Life-18 (QoL-18)
Description: 18-item quality-of-life questionnaire (QoL-18) evaluated a range of participants' behaviors, including mood, engagement, and memory at the end of the study compared to before the use of the MHS. The instrument is scored on a Likert Scale, ranging from 1-5. A higher number indicates better outcome.
Time Frame: The instrument was administered to the participants once -- at the end of their participation in the 6 month study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Gamified Intervention | Non-gamified Intervention
Number analyzed (Participants) | 13 | 15
score on a scale | 3.3 [1 to 5] | 3.6 [1 to 5]

3. Secondary Outcome: 2-item Satisfaction Scale (SS-2)
Description: Quantifies participant's endorsements to two survey questions: How satisfied were they with the MHS? How much progress did they feel like they made? Both questions are scored on a 10-point scale, with a higher value reflecting a better outcome/experience.
Time Frame: The instrument was administered to the participants after the completion of the study duration (i.e., assessed at 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Gamified Intervention | Non-gamified Intervention
Number analyzed (Participants) | 13 | 15
Participants
  Satisfaction: Score of 7 or above | 6 | 9
  Satisfaction: Score of 6 or below | 7 | 6
  Progress: Score of 7 or above | 7 | 10
  Progress: Score of 6 or below | 6 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the study (6 months)
Description: As elaborated in Participant result flow and pre-assignment details, the current study's participant enrollment (and subsequently all reported baseline characteristics, data, and outcomes) only represent the 60 persons living with dementia and do not include nor reflect their respective primary caregivers who assisted in the participant's completion of the study. Following this, adverse event reporting reflect any events that may have occurred that relate to the person living with dementia.
Arm/Group | Gamified Intervention | Non-gamified Intervention
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gamified Intervention (N=30) | Non-gamified Intervention (N=30)
Cancer Treatment (General disorders) | 1 (1) | 0 (0) — Subject's cancer treatment commitments impeded on full participation in study
Seizure (General disorders) | 0 (0) | 1 (1) — Subject reported chronic seizures and requested withdrawal from study due to challenges with fully participating in study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT05422339/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT05422339/ICF_001.pdf